CLINICAL TRIAL: NCT05615584
Title: Multiple Reaction Monitoring (MRM) Versus I 125 Radioimmunoassay (RIA) for the Quantification of Orexin-A/Hypocretin-1 Levels in Cerebrospinal Fluid: a Prospective Diagnostic Validation Study in Patients With Hypersomnolence
Brief Title: Spectrometry (MRM) Versus I 125 Radioimmunoassay (RIA) for Quantification of Orexin-A of Patients With Hypersomnolence
Acronym: MRM-OREX
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RECHMPL22_0072
Record Dates: First submitted 2022-10-26; First posted 2022-11-14 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Narcolepsy; Idiopathic Hypersomnia; Cataplexy
Keywords: orexin/hypocretin; sleepiness
MeSH Terms: conditions — Narcolepsy; Idiopathic Hypersomnia; Cataplexy; Sleepiness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Quantitative mass spectrometry assay — ORX-A determination by quantitative mass spectrometry

SUMMARY:
In humans, selective loss of orexin neurons is responsible for type 1 narcolepsy (NT1), or narcolepsy with cataplexy, or orexin deficiency syndrome.

The International Classification of Sleep Disorders 3rd edition (ICSD-3) distinguishes between hypersomnolence of central origin: NT1, narcolepsy type 2 (NT2), or narcolepsy without cataplexy, and idiopathic hypersomnia (HI). These rare conditions are all characterised by hypersomnolence (excessive daytime sleepiness, or excessive need for sleep), which is the primary and often most disabling symptom. A level of ORX-A in cerebrospinal fluid (CSF) (<110 pg/mL) is a very sensitive and specific biomarker of NT1, currently sufficient for the diagnosis of this condition. In contrast, ORX neurons are thought to be intact in IH and NT2, and the pathophysiological mechanisms underlying these diseases remain unknown. Thus, their diagnosis is based solely on clinical and electrophysiological criteria.

The objective of this project is to determine the validity of a mass spectrometric technique for the determination of ORX-A in the cerebral spinal fluid of patients suffering from hypersomnolence in comparison with the radioimmunoassay which is the reference technique.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 8 years
* Complaint of hypersomnolence and suspected central hypersomnolence
* Benefiting from a standardised assessment: clinical, biological and neurophysiological
* Lumbar puncture necessary for the assessment
* Sufficient cerebrospinal fluid taken for biological analysis (at least 1 ml)
* Signed informed consent

Exclusion Criteria:

* Contraindication to lumbar puncture
* Secondary hypersomnolence
* Refusal to participate in the study or refusal of the lumbar puncture
* Adult protected by law, or subject deprived of liberty, by judicial or administrative decision or patient under guardianship or curatorship
* Subject not affiliated to the French social security system
* Pregnant or breastfeeding woman

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 117 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Orexin-A dosage by Multiple Reaction Monitoring Mass Spectrometry | Day 1 (=day of inclusion)
  Multiple Reaction Monitoring mass spectrometry for orexin-A dosage in cerebrospinal fluid
Orexin-A dosage by radioimmunoassay | Day 1
  Radioimmunoassay for orexin-A dosage in cerebrospinal fluid

SECONDARY OUTCOMES:
Age of onset of hypersomnia symptoms | Day 1
Frequency of cataplexy | Up to 24 hours
Characteristics of cataplexy | Up to 24 hours
Average duration of cataplexy | Up to 24 hours
Epworth sleepiness scale (ESS) | Day 1
  the score will be between 0 and 24, higher scores mean a worse outcome
Narcolepsy severity scale (NSS) | Day 1
  the score will be between 0 and 57, higher scores mean a worse outcome
Hypersomnolence severity scale (IHSS) | Day 1
  the score will be between 0 and 50, higher scores mean a worse outcome
Insomnia severity index | Day 1
  the score will be between 0 and 32, higher scores mean a worse outcome
Iterative sleep latency tests (TILE) | Up to 24 hours
Presence of the HLA allele DQB1*06:02 | Day 1

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No